CLINICAL TRIAL: NCT00280644
Title: Efficacy of Leflunomide on Joint Inflammation and Destruction of Joint Integrity in Active Rheumatoid Arthritis (RA) Patients
Brief Title: Leflunomide in Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HWA486_4022
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Leflunomide

SUMMARY:
Study objectives:

* To provide more insight on the modulation of inflammation and matrix degrading factors in serum and urine by leflunomide in early , active patients with RA and to validate the sensitivity of DEMRI (Dynamic Enhanced Magnetic Resonance Imaging) in detecting inflammatory changes in active RA in response to treatment with leflunomide
* Effect of leflunomide therapy on physical function improvement and Quality of life

ELIGIBILITY:
Inclusion Criteria:

* Patient who has diagnosis of rheumatoid arthritis based upon the ACR (American College of Rheumatology) diagnostic criteria
* Patient who has not ARA functional class IV (ACR 1991 revised criteria). Active disease defined as > 6 swollen or tender joints, by physician and as well as by patient global assessment of disease activity as moderate or worse
* Patient who has active disease defined by a modified Disease Activity Score (DAS)>3.2
* At least one wrist joint with active disease, defined by clinically detectable synovitis at that site due to technical facility of using wrist joint for DEMRI (Dynamic Enhanced Magnetic Resonance Imaging)
* Patient who has received unchanged doses of oral corticosteroids (with a maximum dose of 10 mg prednisone daily or steroid equivalent orally administered ) and concomitant stable doses of nonsteroidal anti-inflammatory drugs for at least 4 weeks before entering the study
* Woman of childbearing potential,who is demonstrated not to be pregnant (by serum pregnancy test) or breast feeding at screening visit, and who is agree to undergo urine pregnancy testing monthly during the study, and serum pregnancy test at the end of the treatment
* Woman of childbearing potential, who agrees to maintain an adequate mean of contraception and not to get pregnant through the study and for 24 months after the discontinuation of the treatment.Man wishing to father a child, who has a consent to discontinue the treatment with study medication, will undergo a drug elimination procedure

Exclusion Criteria:

* The patient who has ARA functional class IV
* The patient who has a history of other inflammatory joint disease, e.g. mixed connective tissue disease, seronegative spondylarthropathy, psoriatic arthritis, Reiter's syndrome, systemic lupus erythematosus, sarcoidosis, history of Felty's syndrome, or any arthritis with onset prior to 16 years of age
* The patient who has a congenital or acquired severe immunodeficiency, a history of cancer or lymphoproliferative disease, or he/she has received total lymphoid irradiation
* The patient who is in known HIV positive status defined by either a positive blood test or clinical diagnosis
* The patient who has been sick with persistent infection or severe infection within 3 months of enrollment
* Known Glucose 6 Phosphate Dehydrogenase (G6PD) deficiency
* The patient who has acute intermittent porphyria
* The patient who has hematopoietic disorder (haemoglobin < 9 g/dl, White Blood Cells < 3500/mm3, platelet count < 120.000/mm3)
* The patient who has impaired coagulation, on treatment with oral anti-coagulants
* The patient who has uncontrolled diabetes, unstable ischaemic heart disease, active inflammatory bowel disease, active peptic ulcer disease or history of active peptic ulcer disease during the previous 4 months (documented by gastroscopy or clinically diagnosed by a physician), recent or history of major traumatic injury, history of malignancy.
* The patient who has clinically relevant cardiovascular, hepatic, neurologic, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult
* Patients body weight is < 45 kg
* The patient who has received therapy within the previous 3 months with any investigational drug, alkylating agents (e.g. cyclophosphamide, chlorambucil), biological agents (e.g. interferon, monoclonal antibodies, growth factor, cytokines).
* The patient who has received other DMARD (Disease Modifying Antirheumatic Drugs) therapy (D-penicillamine, oral or injectable gold, chloroquine, hydroxychloroquine, cyclosporine,MTX) who hasn't been followed by a washout period of 28 days
* Patients who had a therapy of oral corticosteroids exceeding a prednisone equivalent of 10 mg/day, parenteral or intra-articular corticoid injection, within the previous 4 weeks

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-04

PRIMARY OUTCOMES:
The proportion of patients responding according to "28-Joint Disease Activity Score" (DAS28) criteria (a 1.2 point increase compared with pretreatment values), C-Reactive Protein (CRP)

CONTACTS AND LOCATIONS:
Overall Officials: Edibe Taylan, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Istanbul, Turkey (Türkiye)